CLINICAL TRIAL: NCT01879631
Title: Efficacy of Radial Keratotomy in the Optical Rehabilitation of Mild to Moderate Keratoconus Cases
Status: Completed | Type: Observational
Sponsor: Nisa Hastanesi (Other)
Responsible Party: Principal Investigator, Ibrahim Kocak, M.D., Nisa Hastanesi
Other Study IDs: B.30.2.IMU.0.05.05-11; B32IMU0050511 (Other: Istanbul Medipol University clinical trials etics committee)
Record Dates: First submitted 2013-06-11; First posted 2013-06-18 (Estimated); Last update posted 2013-06-18 (Estimated); Status verified 2013-06

CONDITIONS: Radial Keratotomy in Keratoconus Cases
Keywords: radial keratotomy; keratoconus; optical rehabilitation
MeSH Terms: conditions — Keratoconus | interventions — Keratotomy, Radial

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- mild to moderate keratoconus cases: keratoconus with a central corneal thickness (CCT) over 400µm, poor corrected visual acuity (≤0.4 at Snellen visual acuity charts), contact lens intolerance, no apical scarring, no ocular or systemic problem other than keratoconus
  Interventions: Procedure: radial keratotomy

INTERVENTIONS:
Procedure: radial keratotomy

SUMMARY:
Keratoconus is a progressive ectatic disorder that steepens the cornea resulting in a conical shape. Radial Keratotomy can provide an optical rehabilitation by its flattening effect. It can also halt the progression of disease owing to fibrotic activation in perpendicular corneal incisions.

ELIGIBILITY:
Inclusion Criteria:

* keratoconus with a central corneal thickness (CCT) over 400µm,
* poor corrected visual acuity (≤0.4 at Snellen visual acuity charts),
* contact lens intolerance

Exclusion Criteria:

* apical scarring,
* ocular or systemic problem other than keratoconus

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: mild to moderate keratoconus cases
Sampling Method: Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2012-07; Primary Completion 2012-11 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
outcome measures: uncorrected and best spectacle corrected visual acuity, keratometer readings | after surgery - 12 to 52 months
  Preoperative and postoperative uncorrected visual acuity, best spectacle corrected visual acuity, and keratometer readings will be reviewed retrospectively. As reviewed follow up time range is 12 to 52 months, time frame is assessed as " 12 to 52 months"

CONTACTS AND LOCATIONS:
Overall Officials: ibrahim kocak, m.d, Principal Investigator — ophthalmologist
Locations (1):
- Ophthalmology Department, Nisa Hospital, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Result] Utine CA, Bayraktar S, Kaya V, Kucuksumer Y, Eren H, Perente I, Yilmaz OF. Radial keratotomy for the optical rehabilitation of mild to moderate keratoconus: more than 5 years' experience. Eur J Ophthalmol. 2006 May-Jun;16(3):376-84. PMID 16761238